CLINICAL TRIAL: NCT04671485
Title: Randomized, Comparative Pilot Study Evaluating the Effectiveness of autoHYpnosis by Anchoring in the Prevention of Anxiety Related to Wearing the Mask for Radiotherapy of Head and Neck Tumors
Brief Title: Effectiveness of autoHYpnosis in the Prevention of Anxiety During Radiotherapy of Head and Neck Tumors (HYMACO)
Acronym: HYMACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A00813-36
Record Dates: First submitted 2020-12-07; First posted 2020-12-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Tumors
Keywords: Autohypnosis; Anxiety; 5 points Mask; Radiotherapy; Anchoring
MeSH Terms: conditions — Head and Neck Neoplasms; Anxiety Disorders | interventions — Standard of Care; Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM A : standard care (Active Comparator): standard care : Patient undergoing radiotherapy for head and neck tumor with a compression mask, and assessed as anxious about wearing this mask will have standard care
  Interventions: Other: Standard care
- ARM B : standard care + Autohypnosis (Active Comparator): In addition to the standard care, the patient will be called to learn autohypnosis during a specific consultation, with a radiotherapy manipulator trained to learn this technic.
  The patient will use this technic during the centering scanner and the first 5 radiotherapy sessions
  Interventions: Other: Standard care; Other: Autohypnosis
- ARM C : standard care + Musicotherapy (Active Comparator): In addition to the standard care, the patient will choose the music he want to listen from a music database (3 specific moods).
  The chosen music will be broadcast to the patient via a hi-fi system present in the treatment room during the centering scanner and for the first 5 radiotherapy sessions
  Interventions: Other: Standard care; Other: Musicotherapy

INTERVENTIONS:
Other: Standard care — Patient undergoing radiotherapy for head and neck tumor with a compression mask, and assessed as anxious about wearing this mask will have standard care
Other: Autohypnosis — The patient will be called to learn autohypnosis during a specific consultation, with a radiotherapy manipulator trained to learn this technic.
  The patient will use this technic during the centering scanner and the first 5 radiotherapy sessions
  Arms: ARM B : standard care + Autohypnosis
Other: Musicotherapy — the patient will choose the music he want to listen from a music database (3 specific moods).
  The chosen music will be broadcast to the patient via a hi-fi system present in the treatment room during the centering scanner and for the first 5 radiotherapy sessions
  Arms: ARM C : standard care + Musicotherapy

SUMMARY:
HYMACO is a monocentric, randomized comparative pilot study with a total duration of 25 months. The purpose of this study is to evaluate the effectiveness of autoHYpnosis by anchoring in the prevention of anxiety related to wearing the mask for radiotherapy of head and neck tumors.

60 patients will be randomized into 3 arms ARM A : Standard care ARM B : Autohypnosis ARM C : Musicotherapy This study is carried out during the first 5 radiotherapy sessions because this is decisive for the good progress of subsequent sessions

ELIGIBILITY:
Inclusion Criteria:

* Age > or =18
* Patient to receive radiotherapy for a tumor of the head and neck, with a compression mask
* Patient who obtained a score equal to or greater than 56 on the STAI form Y-A questionnaire during the consultation with the radiotherapist before starting treatment
* Patient capable and willing to follow all study procedures in accordance with the protocol
* Patient who understood the study and gave informed consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Contraindication to hypnosis: psychosis, schizophrenia
* Non-French speaking patient
* Significant hearing loss
* Pregnant woman, likely to be, or breastfeeding
* Persons deprived of their liberty or under guardianship (including guardianship)
* Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons
* Patient who has already received radiotherapy to the head or neck with a compression mask

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Anxiety | 5 weeks
  Anxiety will be assessed by the maximum value obtained on the STAI form Y-A questionnaire (state anxiety) on the following 3 measurements: on the centering scanner, at the first and 5th radiotherapy session.

SECONDARY OUTCOMES:
Anxiety | 5 weeks
  Anxiety will also be assessed by a digital rating scale (0 to 10), in the centering or radiotherapy scanner room, just before making the mask before the centering scan and before fitting the mask before each of the first five radiotherapy sessions
Conduct of radiotherapy session | 5 weeks
  The good conduct of the centering scanner and radiotherapy session is determined by:
  * no interruption of the session
  * the absence of vocal intervention by the manipulator during the session
Time required by the hypnopractor for the hypnosis session | 1 hour
  The duration of the conditioning hypnosis session will be collected by the hypnopractor manipulator
Receptivity of patients to hypnosis | 5 weeks
  Corresponds to the time difference in minutes between the actual time of making and wearing the compression mask for the centering scanner and wearing a compression mask for the first 5 radiotherapy sessions and the time estimated by the patient
Assessment of the patient's feelings | 1 hour
  The patient's feelings will be evaluate a questionnaire composed of 5 questions already used in a previous study
Hypnopractic manipulator's satisfaction with the ease of performing the conditioning hypnosis | 1 hour
  Assesing by the hypnopractor manipulator at the end of the session using a digital rating scale (0 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Rémi ETIENNE, Study Chair — Institut de Cancérologie de Lorraine; RENARD Sophie, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France